CLINICAL TRIAL: NCT02218775
Title: A Phase 1 Study of Kappa and Mu Opioid Receptor Occupancy Associated With Repeated Dosing of LY24516302
Brief Title: FASTMAS (Fast-Fail Trials in Mood and Anxiety Spectrum Disorders) Kappa Opioid Receptor Phase 1 Study
Acronym: KOR1
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Funding for the study ended with one subject consented, but not randomized
Sponsor: Andrew Krystal (Other)
Collaborators: Yale University (Other)
Responsible Party: Sponsor-Investigator, Andrew Krystal, Professor, Department of Psychiatry and Behavorial Sciences, Duke University
Organization: Duke University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00052483; HHSN271201200006I (Other: NIMH/NIH)
Record Dates: First submitted 2014-08-15; First posted 2014-08-18 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: Anxiety Disorders
Keywords: Kappa opioid receptor; Mu opioid receptor; LY2456302; Anhedonia; Mood and Anxiety Spectrum Disorders
MeSH Terms: conditions — Anxiety Disorders; Anhedonia | interventions — Aticaprant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LY2456302 (Experimental): LY2456302 dosed orally at 10 mg daily for 2 weeks in healthy volunteers
  Interventions: Drug: LY2456302

INTERVENTIONS:
Drug: LY2456302 — Mood and Anxiety Disorders

SUMMARY:
The available treatments for patients with mood and anxiety spectrum disorders have significant limitations. This study will contribute significantly to public health by taking steps to address these limitations by aiding in the interpretation of a study that: 1) tests a promising new treatment for mood and anxiety spectrum disorders; 2) evaluates a potential target in the brain which could serve as the basis for development of additional new candidate compounds for the treatment of patients with mood and anxiety spectrum disorders; 3) establishes more expeditious methods for evaluating potential new therapies for patients with mood and anxiety spectrum disorders; and 4) specifically establishes methods for the development of new therapies targeting anhedonia, an important RDoC (Research Domain Criteria) endpoint.

DETAILED DESCRIPTION:
This study is an open-label study of two weeks of daily dosing of LY2456302 carried out in 10 healthy volunteers. Subjects will have an initial screening visit where they will have the opportunity to sign informed consent. Those who choose to do so will undergo a series of screening tests to determine whether they meet inclusion/exclusion criteria for this study. Those who qualify will return in 1-7 days for a baseline set of assessments which will include: having MRI imaging carried out on the first day (structural MRI, fMRI during the Monetary Incentive Delay Task, and Resting State Connectivity fMRI), and on the second day having an arterial line placed; undergoing a [11C]-Carfentanil (a synthetic, highly specific mu opioid receptor (mu-OR) agonist) PET mu opioid receptor occupancy study; undergoing a LY2879788 ( radioactive biochemical substance (in particular, a ligand) that is used for diagnosis or for research-oriented study of the receptor systems of the body) PET Kappa Occupancy Study with a single blood sample taken prior to the scan, a sample during the scan, and samples taken at 15, 30, 45, 60, 75, 90, and 120 minutes after the scan to determine whole blood radioactivity, plasma radioactivity, and un-metabolized tracer fraction over time which are needed to determine the input function to the kinetic model for analysis of parameter estimation needed to compute receptor occupancy from the PET scan data; completing a SHAPS; and undergoing a PRT. Note that arterial line placement and serial blood samples are only needed for the LY2879788 scans because, unlike for [11C]-Carfentanil, there is no accepted reference region in the brains of humans for this ligand which necessitates the development of a kinetic model for scan parameter estimation. The next day subjects will begin taking LY2456302 10 mg daily at 11 am and return to the research unit 6 days later for a safety assessment visit. Subjects will then return to the research unit 7 days later during which they will undergo interval history and safety assessments, take their medication at 11 am, and then have MRI imaging at 1:30 pm. A blood sample to determine LY2456302 level will be obtained immediately before and after the MRI imaging session so that we can determine the relationship between ventral striatal activation during the task and serum level of LY2456302. They will then return to the research unit the following day where they will take their last dose of study medication at 11 am and at 1:30 pm will undergo a [11C]-Carfentanil PET mu opioid receptor occupancy study. A blood sample to determine LY2456302 level will be obtained immediately before and after the PET imaging session so that we can determine the relationship between receptor occupancy and serum level of study drug. The following day subjects will have an arterial line placed and undergo LY2879788 PET Kappa Occupancy Study at 9:30 am with a single blood sample taken prior to the scan and samples taken at 15, 30, 45, 60, 75, 90, and 120 minutes after the scan to determine whole blood radioactivity, plasma radioactivity, and un-metabolized tracer fraction over time which are needed to determine the input function to the kinetic model for analysis of parameter estimation needed to compute receptor occupancy from the PET scan data. A blood sample to determine LY2456302 level will also be obtained immediately before and after the PET imaging session so that we can compute the relationship between serum level and receptor occupancy. Subjects will then return 6 days later for a safety assessment after which their participation in the study will end.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 through 65 years of age
* Body mass index 19 through 30 lbs/in2
* Reliable and willing to be available for the duration of the study
* Willing and able to give written informed consent to participate
* Able to understand and comply with instructions
* If female of childbearing potential, must agree to use dual methods of contraception and be willing and able to continue contraception for 6 weeks after the last dose of study drug. Females using oral contraception must have started using it at least 2 months prior to the Baseline Visit
* If male of childbearing potential, must have undergone surgical sterilization (such as a vasectomy) or agree to use a condom used with a spermicide during participation in the study and for 1 month afterward

Exclusion Criteria:

* Any clinically significant abnormality of any of the hematology, clinical, chemistry, or urine drug tests
* Magnetic resonance imaging contraindications at 3 Tesla (e.g., ferromagnetic implants or shrapnel or other incompatibilities)
* Any clinically significant abnormality of the 12-lead ECG; QTc (corrected QT) interval recorded on screening or predose greater than 450 msec
* Any clinically significant history of neurologic disease, cancer, or cardiac, respiratory, metabolic, hepatic, renal, gastrointestinal (except appendectomy), dermatological, venereal, hematological disorder or disease
* Any clinically significant history of Axis I psychiatric disorder, or history of attempted suicide
* History of seeking advice from a physician or counselor for abuse or misuse of alcohol, non-medical drugs, medicinal drugs or other substance abuse, for example, solvents
* Any current or previous recreational use of Class A drugs such as opiates, cocaine, ecstasy, LSD (Lysergic acid diethylamide), and amphetamines (Class B)
* Positive drugs-of-abuse test result at initial exam or at any time during the study
* An alcoholic intake greater than 7 units per week or unwillingness to stop alcohol consumption for the duration of the study {1 unit = 8 g ethanol (250 mL of beer, 1 glass wine [100 mL], 1 measure spirits [30 mL])}
* Use of prescribed medication within 30 days of the first study day, or nonprescription medication including herbal remedies except standard dose vitamin supplements and acetaminophen (up to 4 g/day) within 15 days of the first study drug administration, or any medication that would need to be continued during the study
* Use of any investigational medication within 3 months prior to the start of this study or scheduled to receive an investigational drug other than LY2456302 during the course of this study
* Any smoking of cigarettes or use of any nicotine containing products within the last month or at any time during the study
* History of blood donation in the last 3 months
* History of severe allergies or multiple adverse drug reactions
* Known hypersensitivity to LY2456302
* Any history of a clinically significant gastrointestinal condition
* Any other condition that in the opinion of the investigator would preclude participation in the study
* Pregnant or lactating
* History of peptic ulcer disease or gastritis or positive urea breath test

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-10; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Primary: Kappa opioid receptor occupancy determined with LY2879788 PET imaging; Mu opioid receptor occupancy determined with [11C]-Carfentanil PET imaging | Both on Day 1
  Baseline readings prior to drug dosing
Primary: Kappa opioid receptor occupancy determined with LY2879788 PET imaging; Mu opioid receptor occupancy determined with [11C]-Carfentanil PET imaging | Day 16: Trough LY2879788 PET Kappa Occupancy Study (22.5 hours after dosing)
  KOR occupancy using LY2879788 imaging at time of peak blood level of LY2456302 achieved with 2 weeks of daily dosing of 10 mg. LY2456302.
Peak PET Mu Occupancy | Day 15
  Mu occupancy using [11C]-Carfentanil PET imaging at time of peal blood level of LY2456302 achieved with 2 weeks of daily dosing of 10 mg LY2456302

SECONDARY OUTCOMES:
Reward Circuit Engagement Outcome | Day 0
  Task related fMRI ventral striatal activation occurring with reward and loss anticipation during the Monetary Incentive Delay Task
Reward Circuit Engagement Outcome | Day 14 (time of peak drug level)
  Task related fMRI ventral striatal activation occurring with reward and loss anticipation during the Monetary Incentive Delay Task
Clinical Anhedonia Outcome Utilizing the Snaith-Hamilton Pleasure Scale (SHAPS) | Screening (Day -7 to Day -1)
  The SHAPS is a well validated 14 item questionnaire used to assess anhedonia (the inability to experience pleasure from activities usually found to be enjoyable). Scores on the SHAPS can range from 14 to 56 with higher scores corresponding to higher levels of anhedonia. The SHAPS is the only anhedonia measure to has been found to significantly improve with the administration of a treatment.
Clinical Anhedonia Outcome Utilizing the Snaith-Hamilton Pleasure Scale (SHAPS) | Day 1
  The SHAPS is a well validated 14 item questionnaire used to assess anhedonia (the inability to experience pleasure from activities usually found to be enjoyable). Scores on the SHAPS can range from 14 to 56 with higher scores corresponding to higher levels of anhedonia. The SHAPS is the only anhedonia measure to has been found to significantly improve with the administration of a treatment.
Anhedonia Outcome Utilizing the Snaith-Hamilton Pleasure Scale (SHAPS) | Day 15
  The SHAPS is a well validated 14 item questionnaire used to assess anhedonia (the inability to experience pleasure from activities usually found to be enjoyable). Scores on the SHAPS can range from 14 to 56 with higher scores corresponding to higher levels of anhedonia. The SHAPS is the only anhedonia measure to has been found to significantly improve with the administration of a treatment.
Behavioral Anhedonia Outcome as measured by the Probabilistic Reward Task (PRT) | Day 1
  This outcome measure was designed to objectively assess participants' propensity to modulate behavior as a function of reinforcement history. This task has been validated in multiple independent samples
Behavioral Anhedonia Outcome as measured by the Probabilistic Reward Task (PRT) | Day 15
  Results will be assessed at this time point as compared to Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Andrew D Krystal, MD, MS, Principal Investigator — Duke University
Locations (1):
- Yale University, New Haven, Connecticut, United States

REFERENCES:
- [Background] Rorick-Kehn LM, Witkin JM, Statnick MA, Eberle EL, McKinzie JH, Kahl SD, Forster BM, Wong CJ, Li X, Crile RS, Shaw DB, Sahr AE, Adams BL, Quimby SJ, Diaz N, Jimenez A, Pedregal C, Mitch CH, Knopp KL, Anderson WH, Cramer JW, McKinzie DL. LY2456302 is a novel, potent, orally-bioavailable small molecule kappa-selective antagonist with activity in animal models predictive of efficacy in mood and addictive disorders. Neuropharmacology. 2014 Feb;77:131-44. doi: 10.1016/j.neuropharm.2013.09.021. Epub 2013 Sep 23. PMID 24071566
- [Background] Zheng MQ, Nabulsi N, Kim SJ, Tomasi G, Lin SF, Mitch C, Quimby S, Barth V, Rash K, Masters J, Navarro A, Seest E, Morris ED, Carson RE, Huang Y. Synthesis and evaluation of 11C-LY2795050 as a kappa-opioid receptor antagonist radiotracer for PET imaging. J Nucl Med. 2013 Mar;54(3):455-63. doi: 10.2967/jnumed.112.109512. Epub 2013 Jan 25. PMID 23353688
- [Background] Zheng MQ, Kim SJ, Holden D, Lin SF, Need A, Rash K, Barth V, Mitch C, Navarro A, Kapinos M, Maloney K, Ropchan J, Carson RE, Huang Y. An Improved Antagonist Radiotracer for the kappa-Opioid Receptor: Synthesis and Characterization of (11)C-LY2459989. J Nucl Med. 2014 Jul;55(7):1185-91. doi: 10.2967/jnumed.114.138701. Epub 2014 May 22. PMID 24854795